CLINICAL TRIAL: NCT03640377
Title: Phase II PK/PD Driven Dose Finding Trial of Praziquantel in Children Under Four
Brief Title: Praziquantel in Children Under Age 4
Acronym: PIPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Liverpool (Other); Research Institute for Tropical Medicine, Philippines (Other Government); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Jennifer Friedman, MD, PhD, Director, Center for International Health Research, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 403818
Record Dates: First submitted 2018-07-16; First posted 2018-08-21 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Schistosomiasis; Schistosomiasis Mansoni; Schistosoma Japonicum Infection
MeSH Terms: conditions — Schistosomiasis; Schistosomiasis mansoni; Schistosomiasis japonica | interventions — Praziquantel

STUDY DESIGN:
Intervention Model Description: Children ages 12-48 months who are infected with S. japonicum (Philippines) or S. mansoni (Uganda) will be randomized to receive either 40 or 60 mg/kg of praziquantel at baseline. Six months later, half of each group will receive second treatment at same dose or placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Tablets will be crushed and given with orange juice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Praziquantel 40 mg/kg dose only baseline treatment (Active Comparator): 150 children will receive 40 mg/kg Praziquantel at baseline as single treatment and placebo six months following baseline
  Interventions: Drug: Praziquantel
- Praziquantel 80 mg/kg dose only baseline treatment (Active Comparator): 150 children will receive 80 mg/kg Praziquantel at baseline as single treatment and placebo six months following baseline
  Interventions: Drug: Praziquantel
- Praziquantel 40 mg/kg dose at baseline and 6 months (Active Comparator): 150 children will receive 40 mg/kg Praziquantel at baseline and again six months later.
  Interventions: Drug: Praziquantel
- Praziquantel 80 mg/kg dose at baseline and 6 months (Active Comparator): 150 children will receive 80 mg/kg Praziquantel at baseline and again six months later.
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — Praziquantel given as crushed tablets (40 or 80 mg/kg)

SUMMARY:
The overall goals of this proposal are to conduct a trial to address the significant gaps with respect to our understanding of best approaches to treatment of children ages 1-4 with intestinal schistosomiasis. Over 200 million individuals worldwide are infected with one of three predominant species of schistosomes, with over half of infections occurring in children. Recent studies have highlighted the fact that many children experience first infections before the age of two, with the prevalence of infection among children under four mirroring the prevalence of older children from the same community. Importantly, praziquantel (PZQ), the drug used worldwide for the treatment of schistosomiasis, is only FDA approved among adults and children over the age of four. Only one small study led by co-PI Bustinduy has evaluated the pharmacokinetic/pharmacodynamics (PK/PD) of PZQ in children. That study, conducted among children ages 3-8, strongly suggests that the current dose of 40 mg/kg is insufficient, with lower cure rates than found at 60 mg/kg.

In endemic settings, PZQ is most often administered as part of school based, or community wide preventive chemotherapy campaigns. Currently, none of the 28 schistosomiasis endemic African nations or The Philippines includes children under the age of four in control programs. The reasons for this are multifactorial and include a) lack of sufficient PK/PD data in this age group, with none in children under three, b) lack of safety data at a dose of 80 mg/kg, c) lack of data addressing the impact of treatment on key growth and nutritional outcomes in this vulnerable age group hampering prioritization of treatment, d) no PK/PD studies conducted in the context of pediatric S. japonicum and e) FDA labeling that does not include young children.

The goals of this proposal are to conduct a randomized, controlled Phase II trial to be conducted in an S. mansoni endemic region of Uganda and an S. japonicum endemic region of The Philippines with N=600 children ages 1-4, that will address many of the current gaps that are hindering treatment of young children. Specifically in SA1 we will 1) assess PK/PD of PZQ dosing among children under the age of 4 at doses of 40 versus 80 mg/kg, 2) expand PD endpoints to include state of the art antigen tests and morbidity outcomes, 3) assess the PK/PD of both PZQ enantiomers, and 4) address the innovative hypothesis that environmental enteropathy (EE) contributes to the significant inter-individual variability observed in PZQ PK/PD. In SA2, we will 1) assess the safety of PZQ administered at 80 mg/kg in two large cohorts of very young children, 2) assess the impact of two different treatment intervals (6 vs 12 months) on nutritional status, growth, and anemia risk, and 3) address innovative hypotheses regarding mechanisms through which schistosomiasis contributes to morbidity in this age group including EE and gut microbial translocation with consequent systemic immune activation.

DETAILED DESCRIPTION:
Over 200 million individuals worldwide are infected with one of three predominant species of schistosomes, with over half of infections occurring in children.1 Recent studies have highlighted the fact that many children experience their first infections before the age of two, with the prevalence of infection among children under four mirroring the prevalence of older children and adults from the same community.2 Importantly, schistosomiasis has been implicated as a cause of linear growth stunting, undernutrition, anemia, and deficits in neurodevelopment among children over the age of four, representing a significant proportion of the global burden of disease due to schistosomiasis.3 Little is known with respect to the impact of schistosomiasis on key morbidities among the highly vulnerable group of children under four.

In the 1980s, Praziquantel (PZQ) was approved for the treatment of schistosomiasis among adults and children ages four and older, and remains FDA approved only for this age group. In 2008, the WHO funded studies to address the safety and parasitologic efficacy of PZQ in the context of S. haematobium and S. mansoni in young children. Based on these and other studies, the WHO in 2011 issued a report recommending that pre-school age children be treated as part of "regular health services."4 This recommendation was based on studies that did not a) evaluate pharmaco-kinetics/dynamics (PK-PD) in this age group, b) evaluate parasitologic efficacy in S. japonicum or c) evaluate the impact of treatment on key schistosomiasis-related morbidities. Since that time, co-PI Bustinduy led the first study of the PK-PD of PZQ at both 40 and 60 mg/kg dosing among children ages 3-8. Results from that study, albeit small, showed that higher doses are likely needed, particularly for younger children. Authors urged further study of higher doses in this age group, the causes of the significant inter-subject variability in PK-PD, better PD indices linking drug exposure to treatment effects, and enantiomer activity across all three species before introduction of monoenantiomeric formulations.5

Thus, significant lacunae remain with respect to treatment of pre-school age children, which contribute to the persistent exclusion of this vulnerable age group from preventive chemotherapy campaigns, with none of the 28 schistosomiasis endemic African nations or The Philippines currently including children under the age of four in control programs.2 In this application, we propose a trial to investigate the off label use of PZQ in children under the age of four. The trial will be conducted at two sites, with high prevalence of intestinal schistosomiasis due to S. mansoni (Uganda) and S. japonicum (The Philippines) employing a two arm single blind, placebo controlled modified cross-over trial design among N=600 children ages 1-4. Children who are infected with schistosomiasis will be randomized at baseline to receive 40 or 80 mg/kg of PZQ. At six months, we will re-randomize half of each baseline group to receive a treatment at the same dose or placebo. This will allow us to evaluate the impact of 6 versus 12 month treatment intervals on key measures of morbidity which, importantly, will inform frequency of treatment needed in this young age group. Successful execution of the following specific aims for this trial will address the significant aforementioned gaps:

SA1 To assess the PK/PD of PZQ administered at different dose regimens. SA1a To measure drug efficacy as per standard parasitological endpoints (Cure Rate and Egg Reduction Rate) at 4 +/- 1 weeks post-PZQ.

SA1b To expand PD endpoints for drug efficacy to include state-of-the art antigen tests to accurately capture residual worm burden (Circulating Cathodic and Anodic Antigens (CCA and CAA)).

SA1c To evaluate the PK/PD of both PZQ enantiomers given the concern that this varies across species and has varied in studies of S. mansoni.

SA1d To assess the role of environmental enteropathy in inter-individual variability in PZQ area under the curve (AUC) demonstrated in this age group.

SA2 To assess the safety and impact of PZQ treatment (dose and interval) on key measures of morbidity 6 and 12 months after initial treatment and mechanisms mediating morbidity.

SA2a To further evaluate the safety of higher PZQ dosing (60 mg/kg), particularly among the unstudied group of very young children ages 1-2.

SA2b To evaluate the impact of different doses (40 vs. 80 mg/kg) and varying dosing intervals (every 6 or 12 months) on iron status, hemoglobin, and age and gender adjusted longitudinal growth and nutritional status as captured by height and weight for age, and weight for height z-scores as determined by WHO Anthro.

SA2c To evaluate the mechanistic role of environmental enteropathy (EE) in the pathogenesis of schistosomiasis related morbidities. We will capture state of the art biomarkers of EE including fecal calprotectin, urine lactulose:mannitol ratio, serum endotoxin, serum endotoxin core antibody, and pro-inflammatory cytokines and employ Path Modeling techniques to identify mechanistic pathways.

ELIGIBILITY:
Inclusion Criteria:

* S. japonicum or S. mansoni infection by urine CCA
* Otherwise healthy as determined by history and physical examination conducted by the study physician at the second stage screening
* Age 12-48 months inclusive
* Parental consent to participate.

Exclusion Criteria:

* Parental inability to provide informed consent
* Significant disease/illness as determined by history or physical exam. This includes a severe acute illness or chronic disease as defined by greater than 3 months duration and significantly impacting a child's daily activities.
* Severe wasting as defined by WHZ < -3,
* Severe anemia (hemoglobin < 7 g/dL)
* Exposure to immuno-modulatory therapeutics.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | Four weeks post treatment
  Treatment efficacy as captured by egg reduction rate
Treatment efficacy | Four weeks post treatment
  Treatment efficacy as captured by cure rate

SECONDARY OUTCOMES:
Iron status | Six and 12 months following treatment
  Assess impact of varying doses and frequency of dosing on iron status
Hemoglobin | Six and 12 months following treatment
  Assess impact of varying doses and frequency of dosing on hemoglobin
Age and gender adjusted linear growth | Six and 12 months following treatment
  Assess impact of varying doses and frequency of dosing on linear growth
Age and gender adjusted nutritional status | Six and 12 months following treatment
  Assess impact of varying doses and frequency of dosing on nutritional status
Biomarker of inflammation-CRP | Six and 12 months following treatment
  CRP
Biomarker of inflammation-IL-6 | Six and 12 months following treatment
  serum IL-6
Biomarker of inflammation-TNF-alpha | Six and 12 months following treatment
  serum TNF-alpha
Fecal Calprotectin | Six and 12 months following treatment
  A measure of gut inflammation
Urine Lactulose-Mannitol Ratio | 12 months following treatment
  A measure of environmental enteropathy

OTHER OUTCOMES:
Pharmacokinetic profile of Praziquantel | up to 24 hours post treatment
  Area under the curve will be measured at discrete intervals from time 0 to 24 hours following treatment
Pharmacokinetic profile of Praziquantel | up to 24 hours post treatment
  Maximum plasma concentration (CMax) will be captured by measure Praziquantel at discrete intervals from time 0 to 24 hours following treatment
Pharmacodynamic profile of Praziquantel | 4 weeks post treatment
  The number of participants who achieve an egg reduction rate of 90% or greater
Pharmacodynamic profile of Praziquantel | 4 weeks post treatment
  The number of participants who achieve complete cure as defined by 0 eggs per gram of feces at 4 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Medical Research Council, Entebbe, Uganda
- London School of Tropical Hygiene and Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from the trial will be made available to interested investigators following IRB approval to provide these de-identified data. Specifically, after research data set has been cleaned, finalized, and all identifiers removed, the PIs will provide timely release and sharing of the final research data for use by other researchers. In addition, this study will generate samples collected young children. Upon discussion with the Principal Investigators and based on availability of samples, residual stored samples may be shared following IRB approval to provide these de-identified samples to interested researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year of trial completion and up to five years after.

REFERENCES:
- [Derived] Bustinduy AL, Edielu A, Ayebazibwe GK, Nakyesige R, Anguajibi V, Mpooya S, Nassuna J, Adriko M, Elliott A, van Dam G, Corstjens P, Pach S, Wu H, Colt S, Mawa PA, Muheki E, Kabatereine NB, Webb EL, Friedman JF. Safety and efficacy of praziquantel 40 mg/kg versus 80 mg/kg in preschool-aged children with intestinal schistosomiasis in Uganda: a 2 x 2 factorial, double-blind, placebo-controlled, phase 2 randomised trial. Lancet Glob Health. 2025 Jun;13(6):e1091-e1100. doi: 10.1016/S2214-109X(25)00095-6. PMID 40412398
- [Derived] Webb EL, Edielu A, Wu HW, Kabatereine NB, Tukahebwa EM, Mubangizi A, Adriko M, Elliott AM, Hope WW, Mawa PA, Friedman JF, Bustinduy AL. The praziquantel in preschoolers (PIP) trial: study protocol for a phase II PK/PD-driven randomised controlled trial of praziquantel in children under 4 years of age. Trials. 2021 Sep 6;22(1):601. doi: 10.1186/s13063-021-05558-1. PMID 34488846